CLINICAL TRIAL: NCT07284537
Title: Pioneering Video-Based Neurocritical Care Education in Palestine: A Randomized Controlled Trial on Nursing Students' Knowledge, Attitude, Practice, and Self-Confidence Toward External Ventricular Drainage
Brief Title: Neurocritical Care Video Training in Palestine: RCT on Nursing Students' EVD Knowledge, Attitude, Skills, Confidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modern University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: muc026\2025
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Clinical Competence; Self-Confidence; Knowledge Level
Keywords: Neurocritical Care Skills; Clinical Competence; Confidence; Nursing Education; knowledge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- class a (Experimental): Video based education
  Interventions: Other: video based education
- class b (Placebo Comparator): flashcards
  Interventions: Other: Flashcard

INTERVENTIONS:
Other: video based education — Participants assigned to this arm will attend a 57-minute classroom session consisting of a prerecorded instructional video covering essential concepts related to external ventricular drainage (EVD). The session will be delivered once, in a group format, using a classroom projector. No additional materials or activities will be provided during the session.
  Arms: class a
Other: Flashcard — Participants in this arm will receive a single 57-minute classroom session using printed or digital flashcards containing EVD-related theoretical content. Participants will review the flashcards individually under supervision. This group will not view any video material during the session, and no audiovisual resources will be provided.
  Arms: class b

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a video-based educational program on nursing students' knowledge, attitude, self-reported practice, and confidence related to external ventricular drainage (EVD) care. The study will be conducted among third- and fourth-year undergraduate nursing students enrolled in the critical care course at Modern University College, West Bank, Palestine. Participants will be randomly assigned in a 1:1 ratio to either a structured 57-minute video-based educational session or an equivalent flashcard-based session covering the same content. All participants will complete pre- and post-intervention assessments to measure changes in EVD-related knowledge, attitude, self-reported practice, and confidence.

DETAILED DESCRIPTION:
This single-center, single-blind randomized controlled trial is designed to compare two educational methods-video-based instruction and flashcard-based theoretical learning-among undergraduate nursing students. The purpose of the study is to examine whether a structured video-based educational session influences students' knowledge, attitude, self-reported practice, and confidence in relation to external ventricular drainage (EVD) care.

Participants will be recruited from third- and fourth-year nursing students enrolled in the critical care course who have not yet completed the neurological nursing module. Eligible students must be actively enrolled in the course, willing to participate, and able to complete all study procedures. Students with prior formal EVD training or clinical exposure to EVD care will be excluded.

A simple randomization procedure will assign participants to either the video-based education group or the flashcard-based education group. Allocation concealment will be maintained using sealed, opaque envelopes prepared by an independent researcher. Participants will be blinded to the specific intervention under investigation, and outcome assessors will be unaware of group assignments.

Interventions

Video-Based Education Group:

Participants will view a 57-minute instructional video covering essential concepts related to EVD, including indications, monitoring principles, equipment, procedures, and safety considerations. The session will be delivered in a classroom setting, and the content will align with standard neurocritical care educational materials.

Flashcard-Based Education Group:

Participants assigned to the control group will review a set of illustrated flashcards containing the same educational content presented in the video. The flashcard session will match the duration of the video-based session and will provide a structured, text-based theoretical review.

To minimize contamination, both sessions will be delivered separately on the same day in different classrooms. Access to materials will be restricted until data collection is completed.

Data Collection

Pre-intervention assessments will be administered immediately before the educational sessions, and post-intervention assessments will be collected immediately afterward. The assessment tool includes demographic questions and structured items measuring EVD-related knowledge, attitude, self-reported practice, and subjective confidence.

All data will be collected electronically using secure online forms. Responses will be coded to maintain confidentiality, and group labels will not be visible to the assessors evaluating completed questionnaires.

Data Analysis

Data will be analyzed using descriptive and inferential statistics as planned in the study protocol. Analyses will include comparisons of pre- and post-intervention scores within and between groups, as well as appropriate statistical modeling to adjust for baseline differences. A significance threshold of 0.05 will be used.

Ethical Considerations

Ethical approval was obtained from the institutional research ethics committee. Participation is voluntary, and informed consent will be obtained electronically. Confidentiality will be maintained by assigning coded identifiers, and data will be stored securely. Both groups will receive access to all educational materials after data collection is completed.

ELIGIBILITY:
Inclusion Criteria:

* students registered at MUC, such as 3rd and 4th year

Exclusion Criteria:

* students in 1st and 2nd year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Knowledge Score Measured by the EVD Knowledge Questionnaire | Baseline (pre-test) and immediately after the intervention (post-test)
  Description:
  Knowledge about external ventricular drainage will be assessed using an 11-item multiple-choice questionnaire. Each correct answer receives 1 point and each incorrect answer receives 0, yielding a total score of 0-11. Higher scores indicate greater knowledge.
  Unit of Measure:
  Score (0-11)
Self-Confidence Visual Analog Scale (VAS) | Baseline (pre-test) and immediately after the intervention (post-test)
  Self-confidence in performing EVD-related procedures will be measured using a 10-point visual analog scale (VAS), where 0 indicates no confidence and 10 indicates maximum confidence.
  Unit of Measure: Score (0-10)
Attitude Score Measured by the EVD Attitude Scale | At baseline and immediately after completion of the intervention
  Description:
  Attitude toward EVD care will be measured using a 6-item Likert scale from 1 (strongly disagree) to 5 (strongly agree), producing a total score of 6-30. Higher scores represent more positive attitudes.
  Unit of Measure:
  Score (6-30)
EVD Practice Checklist | Baseline (pre-test) and immediately after the intervention (post-test)
  Practical EVD skills will be evaluated using a standardized 10-item EVD Practice Checklist. Each item is marked as completed (1) or not completed (0), producing a total score from 0 to 10, which is converted into a percentage. Higher percentages indicate better EVD practice performance.
  Unit of Measure: Percentage (points)

CONTACTS AND LOCATIONS:
Overall Officials: Nawaf Raed Amro, Master Degree, Study Director — Modern University College
Locations (1):
- Modern University College, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Google scholar Profile — https://scholar.google.com/citations?user=8CgLuXUAAAAJ&hl=ar&oi=ao

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT07284537/Prot_SAP_000.pdf